CLINICAL TRIAL: NCT00843024
Title: TXA107979: A Randomized, Multicenter, Placebo-Controlled, Parallel Group Study to Evaluate the Efficacy and Safety of a Combination Product Containing Sumatriptan and Naproxen Sodium for the Acute Treatment of Migraine in Adolescents
Brief Title: Migraine Study in Adolescent Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 107979
Record Dates: First submitted 2009-02-12; First posted 2009-02-13 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2016-11

CONDITIONS: Migraine Disorders
Keywords: Migraine with or without aura; Migraine efficacy; Migraine; Migraine headache; Adolescent migraine; TREXIMET; Sumatriptan succinate; Naproxen sodium; Migraine, acute
MeSH Terms: conditions — Migraine Disorders | interventions — Sumatriptan; Naproxen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sumatriptan and Naproxen 1 (Experimental): Sumatriptan succinate and naproxen sodium combination 10mg/60mg
  Interventions: Drug: Sumatriptan and Naproxen Sodium
- Sumatriptan and Naproxen 2 (Experimental): Sumatriptan succinate and naproxen sodium combination 30mg/180mg
  Interventions: Drug: Sumatriptan and Naproxen Sodium
- Sumatriptan and Naproxen 3 (Experimental): Sumatriptan succinate and naproxen sodium combination 85mg/500mg
  Interventions: Drug: Sumatriptan and Naproxen Sodium
- Placebo (Placebo Comparator): Placebo to match
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sumatriptan and Naproxen Sodium — Sumatriptan succinate and naproxen sodium
  Arms: Sumatriptan and Naproxen 1; Sumatriptan and Naproxen 2; Sumatriptan and Naproxen 3
Drug: Placebo — Placebo to match
  Arms: Placebo

SUMMARY:
This study was designed to determine how well the combination medication, sumatriptan and naproxen sodium, treats migraine headache in adolescents 12-17 years old

DETAILED DESCRIPTION:
The purpose of this study is to determine whether the combination product, sumatriptan and naproxen sodium, is effective compared to placebo in the treatment of acute migraine in adolescent subjects 12-17 years old. Subjects will treat two migraine attacks over a ~25 week period.

ELIGIBILITY:
Inclusion Criteria: Subjects eligible for enrollment in the study must meet all of the following criteria:

1. Subject is >/=12 years of age and </=17 years of age at the Screening Visit.
2. Subject has migraine with or without aura (ICHD-II criteria, 1.2.1 or 1.1). A history of at least two, but no more than eight attacks per month, for the six months prior to the Screening Visit is required. Attacks should last a minimum of three hours and be associated with moderate-to-severe headache pain.
3. Subject is able to distinguish migraine from other headaches (i.e., tension-type headaches).
4. Male or female subjects. Female subjects are eligible for participation in the study if they are:

   1. Females of non-childbearing potential; or
   2. Females of childbearing potential, and who have a negative urine pregnancy test at screening, and agree to use one of the GlaxoSmithKline (GSK)-specified highly effective methods for avoiding pregnancy
5. Any subject taking oral contraceptives at enrollment must be on a stable regimen for at least 2 months prior to screening.
6. Subject and subject's parent or legal guardian are able to read and write English or Spanish.
7. Subject is able to read, comprehend, and complete subject diaries.
8. Subject's parent or legal guardian is willing and able to provide Informed Consent prior to subject entry into the study.
9. Subject is willing and able to provide Informed Assent prior to entry into the study (if required).

   -

Exclusion Criteria:

* Subjects meeting any of the following criteria must not be enrolled in the study:

  1. Subject is < 74 pounds (33.3 kg).
  2. Subject has ≥15 headache days per month in total (migraine, probable migraine, or tension-type), retinal (ICHD-II 1.4), basilar (ICHD-II 1.2.6), or hemiplegic migraine (ICHD-II 1.2.4), or secondary headaches.
  3. Subject, in the investigator's opinion is likely to have unrecognized cardiovascular or cerebrovascular disease.
  4. Subject has uncontrolled hypertension at screening or is taking any angiotensin-converting enzyme (ACE) inhibitor or angiotensin receptor blocker.
  5. Subject has a history of congenital heart disease, cardiac arrhythmias requiring medication, or a history of a clinically significant electrocardiogram abnormality that, in the investigator's opinion, contraindicates participation in this study.
  6. Subject has evidence or history of any ischemic vascular diseases including: ischemic heart disease, ischemic abdominal syndromes, peripheral vascular disease, or signs/symptoms consistent with any of the above.
  7. Subject has evidence or history of central nervous system pathology including stroke and/or transient ischemic attacks (TIAs), epilepsy or structural brain lesions which lower the convulsive threshold, or has been treated with an antiepileptic drug for seizure control within 5 years prior to screening.
  8. Subject has a history of impaired hepatic or renal function that, in the investigator's opinion, contraindicates participation in this study.
  9. Subject has hypersensitivity, allergy, intolerance, or contraindication to the use of any triptan, NSAID, or aspirin (including all sumatriptan and naproxen preparations) or has nasal polyps and asthma.
  10. Subject has used an ergot medication in the previous three months for migraine prophylaxis or is taking a medication that is not stabilized (i.e., change of dose within the past 2 months) for either chronic or intermittent migraine prophylaxis or for a co-morbid condition that is not stabilized.
  11. Subject has a recent history of regular use of opioids or barbiturates for treatment of their migraine headache and/or other non-migraine pain. Regular use is defined as an average of 4 days per month over the last 6 months.
  12. Subject has taken, or plans to take, a monoamine oxidase inhibitor (MAOI), including herbal preparations containing St. John's Wort (Hypericum perforatum), anytime within the two weeks prior to screening through two weeks post treatment.
  13. Subject has a history of any bleeding disorder or is currently taking any anti-coagulant or any antiplatelet agent.
  14. Subject has evidence or history of any gastrointestinal surgery, GI ulceration, or perforation in the past six months, gastrointestinal bleeding in the past year, or evidence or history of inflammatory bowel disease.
  15. Subject is pregnant, actively trying to become pregnant, or breast feeding or subject is not willing to have pregnancy test(s).
  16. Subject tests positive for illicit substances on toxicology screen, or has evidence of alcohol or substance abuse within the last year, or any concurrent medical or psychiatric condition which, in the investigator's judgment, will likely interfere with the study conduct, subject cooperation, or evaluation and interpretation of the study results, or which otherwise contraindicates participation in this clinical trial.
  17. Subject has participated in any investigational drug trial within the previous 4 weeks or plans to participate in another study at any time during this study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 589 (Actual)
Dates: Start 2008-12; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (74):
- United States (74):
  - GSK Investigational Site, Gilbert, Arizona
  - GSK Investigational Site, Litchfield Park, Arizona
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Conway, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Chico, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Fullteron, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Roseville, California
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Santa Monica, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Fairfield, Connecticut
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pensacola, Florida
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Savannah, Georgia
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Oak Lawn, Illinois
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Anderson, Indiana
  - GSK Investigational Site, Terre Haute, Indiana
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Wichita, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Lexington, Kentucky
  - GSK Investigational Site, Pikesville, Maryland
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Vorhees, New Jersey
  - GSK Investigational Site, Willingboro, New Jersey
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Amherst, New York
  - GSK Investigational Site, Mineola, New York
  - GSK Investigational Site, Mount Vernon, New York
  - GSK Investigational Site, Schenectady, New York
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, West Chester, Ohio
  - GSK Investigational Site, Westerville, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Salem, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Simpsonville, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Clarksville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Seattle, Washington
  - GSK Investigational Site, Vancouver, Washington
  - GSK Investigational Site, Wenatchee, Washington
  - GSK Investigational Site, Madison, Wisconsin
  - GSK Investigational Site, Middleton, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Brandes JL, Kudrow D, Stark SR, O'Carroll CP, Adelman JU, O'Donnell FJ, Alexander WJ, Spruill SE, Barrett PS, Lener SE. Sumatriptan-naproxen for acute treatment of migraine: a randomized trial. JAMA. 2007 Apr 4;297(13):1443-54. doi: 10.1001/jama.297.13.1443. PMID 17405970
- [Derived] Derosier FJ, Lewis D, Hershey AD, Winner PK, Pearlman E, Rothner AD, Linder SL, Goodman DK, Jimenez TB, Granberry WK, Runken MC. Randomized trial of sumatriptan and naproxen sodium combination in adolescent migraine. Pediatrics. 2012 Jun;129(6):e1411-20. doi: 10.1542/peds.2011-2455. Epub 2012 May 14. PMID 22585767
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107979 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- 12 to 14 Years Age Group: Single-blind Phase: Participants 12 to 14 years old treated one moderate to severe migraine attack with one tablet of single-blind placebo within a 12-week period. After completion of the run-in phase, participants were randomized to one of four double-blind treatment groups.
- 15 to 17 Years Age Group: Single-blind Phase: Participants 15 to 17 years old treated one moderate to severe migraine attack with one tablet of single-blind placebo within a 12-week period. After completion of the run-in phase, participants were randomized to one of four double-blind treatment groups.
- Placebo: After completing the single-blind phase, participants received a single matching placebo tablet taken within a 12-week period
- Sumatriptan 10 mg/ Naproxen 60 mg: After completing the single-blind phase, participants received a single combination tablet of sumatriptan 10 milligrams (mg) and naproxen sodium 60 mg taken within a 12-week period
- Sumatriptan 30 mg/ Naproxen 180 mg: After completing the single-blind phase, participants received a single combination tablet of sumatriptan 30 mg and naproxen sodium 180 mg taken within a 12-week period
- Sumatriptan 85 mg/ Naproxen 500 mg: After completing the single-blind phase, participants received a single combination tablet of sumatriptan 85 mg and naproxen sodium 500 mg taken within a 12-week period
Period: Single-blind Placebo Run-In Phase
Arm/Group | 12 to 14 Years Age Group: Single-blind Phase | 15 to 17 Years Age Group: Single-blind Phase | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Started | 408 | 457 | 0 | 0 | 0 | 0
Completed | 268 | 321 | 0 | 0 | 0 | 0
Not Completed | 140 | 136 | 0 | 0 | 0 | 0
Not completed — Did not meet continuation criteria | 79 | 74 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 36 | 31 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 19 | 18 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 5 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 0 | 1 | 0 | 0 | 0 | 0
Period: Double-blind Treatment Phase
Arm/Group | 12 to 14 Years Age Group: Single-blind Phase | 15 to 17 Years Age Group: Single-blind Phase | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Started | 0 | 0 | 176 | 119 | 117 | 177
Completed | 0 | 0 | 145 | 96 | 97 | 152
Not Completed | 0 | 0 | 31 | 23 | 20 | 25
Not completed — No opportunity to treat migraine | 0 | 0 | 20 | 10 | 13 | 14
Not completed — Lost to Follow-up | 0 | 0 | 8 | 4 | 4 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 6 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 3 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 3 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: A single matching placebo tablet taken within a 12-week period
- Sumatriptan 10 mg/ Naproxen 60 mg: A single combination tablet of sumatriptan 10 milligrams (mg) and naproxen sodium 60 mg taken within a 12-week period
- Sumatriptan 30 mg/ Naproxen 180 mg: A single combination tablet of sumatriptan 30 mg and naproxen sodium 180 mg taken within a 12-week period
- Sumatriptan 85 mg/ Naproxen 500 mg: A single combination tablet of sumatriptan 85 mg and naproxen sodium 500 mg taken within a 12-week period
- Total: Total of all reporting groups
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg | Total
Number analyzed (Participants) | 145 | 96 | 97 | 152 | 490
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics are provided for participants in the Intent-to-Treat (ITT) Population, comprised of all participants who provided any post-treatment efficacy assessment.
  Years | 14.7 (1.76) | 14.8 (1.81) | 14.7 (1.65) | 14.8 (1.69) | 14.7 (1.72)
Gender [Count of Participants; unit: Participants]
  Female | 85 | 52 | 56 | 94 | 287
  Male | 60 | 44 | 41 | 58 | 203
Race/Ethnicity, Customized [Number; unit: participants]
  African American/African Heritage | 25 | 17 | 9 | 12 | 63
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 1 | 0 | 0 | 3 | 4
  Native Hawaiian or other Pacific Islander | 1 | 0 | 0 | 0 | 1
  White | 108 | 75 | 84 | 130 | 397
  African American/African Heritage and White | 2 | 1 | 1 | 2 | 6
  American Indian or Alaska Native and White | 1 | 2 | 2 | 3 | 8
  Asian and Native Hawaiian/other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Asian and White | 3 | 1 | 0 | 1 | 5
  Native Hawaiian/ other Pacific Islander and White | 1 | 0 | 1 | 0 | 2
  Missing | 2 | 0 | 0 | 0 | 2
Weight [Mean (Standard Deviation); unit: Kilograms (kg)] | 63.8 (16.67) | 64.2 (19.29) | 62.8 (14.49) | 66.8 (19.13) | 64.6 (17.63)
Body Mass Index [Mean (Standard Deviation); unit: Kilograms per meters squared (kg/m^2)] — Body Mass Index is calculated as: weight (kg)/height (m^2)
  Kilograms per meters squared (kg/m^2) | 23.5 (5.28) | 23.3 (5.62) | 22.9 (4.53) | 24.6 (5.68) | 23.7 (5.36)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Pain Free at 2 Hours Post-dose
Description: Participants were evaluated (self-assessment) for pain intensity by using a 4-point rating scale: 0=none, 1=mild, 2=moderate, and 3=severe. Participants with pain-free response were considered as those who had a reduction in migraine headache pain from moderate (score=2) or severe (score=3) at baseline to none (score=0) post-treatment, without the use of rescue medication (additional medication taken by participants for the treatment of migraine pain or associated symptoms) prior to or at 2 hours post-dose.
Time Frame: 2 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: ITT Population: participants who took a dose of double-blind randomized treatment and provided some assessment of their migraine pain or associated symptoms. Participants were not included in this analysis if their baseline pain was not moderate or severe, or if they had no post-baseline evaluation of pain up to the time point analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 142 | 96 | 97 | 150
participants
  Total Population, n=142, 96, 97, 150 | 14 | 28 | 26 | 36
  12-14 years, n=70, 43, 46, 65 | 10 | 18 | 13 | 17
  15-17 years, n=72, 53, 51, 85 | 4 | 10 | 13 | 19
Statistical Analysis 1: Comparison: Placebo vs Sumatriptan 10 mg/ Naproxen 60 mg; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — Adjusted for multiplicity according to the fixed sequence testing strategy; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.09 to 0.30] — Sumatriptan 10 mg/Naproxen 60 mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Sumatriptan 30 mg/ Naproxen 180 mg; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — Adjusted for multiplicity according to the fixed-sequence testing strategy; Mean Difference (Final Values) = 0.16, 95% CI 2-sided [0.07 to 0.26] — Sumatriptan 30 mg/Naproxen180 mg minus placebo
Statistical Analysis 3: Comparison: Placebo vs Sumatriptan 85 mg/ Naproxen 500 mg; Test type: Superiority or Other; p = 0.003, Cochran-Mantel-Haenszel — Adjusted for multiplicity according to the fixed-sequence testing strategy; Mean Difference (Final Values) = 0.13, 95% CI 2-sided [0.05 to 0.22] — Sumatriptan 85 mg/Naproxen 500 mg minus placebo

2. Secondary Outcome: Number of Participants Sustained Pain-free From 2-24 Hours
Description: Participants with sustained pain-freedom were defined as those with pain-freedom at 2 hours post-dose that was maintained up to 24 hours post-treatment without the use of rescue medication.
Time Frame: 2 to 24 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: ITT Population. Participants were not included in pain-related analyses if their baseline pain was not moderate or severe, and were not included in analyses of pain or symptoms if they had no post-baseline evaluation of the relevant pain or symptom up to the time point analyzed.
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 142 | 96 | 97 | 150
participants
  Total Population, n=142, 96, 97, 150 | 13 | 23 | 24 | 35
  12-14 years, n=70, 43, 46, 65 | 10 | 14 | 12 | 17
  15-17 years, n=72, 53, 51, 85 | 3 | 9 | 12 | 18

3. Secondary Outcome: Number of Participants Photophobia-free at 2 Hours Post-dose
Description: The number of participants who did not have photophobia (sensitivity to light) at 2 hours post dose was analyzed.
Time Frame: 2 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 144 | 96 | 96 | 151
participants
  Total Population, n=144, 96, 96, 151 | 59 | 57 | 47 | 89
  12-14 years, n=71, 43, 46, 65 | 33 | 29 | 24 | 41
  15-17 years, n=73, 53, 50, 86 | 26 | 28 | 23 | 48

4. Secondary Outcome: Number of Participants Phonophobia-free at 2 Hours Post-dose
Description: The number of participants who did not have phonophobia (sensitivity to sound) at 2 hours post dose was analzyed.
Time Frame: 2 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 144 | 96 | 96 | 151
participants
  Total Population, n=144, 96, 96, 151 | 60 | 59 | 55 | 90
  12-14 years, n=71, 43, 46, 65 | 34 | 32 | 33 | 41
  15-17 years, n=73, 53, 50, 86 | 26 | 47 | 22 | 49

5. Secondary Outcome: Number of Participants Pain-free at 1 Hour Post-dose
Description: Participants with a pain-free response at 1 hour post-dose were considered as those who had a reduction in migraine headache pain from moderate (a score of 2) or severe (a score of 3) at baseline to none (a score of 0) post-treatment, without the use of rescue medication prior to or at 1 hour post dose.
Time Frame: 1 hour after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 142 | 96 | 97 | 150
participants
  Total Population, n=142, 96, 97, 150 | 6 | 9 | 6 | 11
  12-14 years, n=70, 43, 46, 65 | 4 | 7 | 2 | 4
  15-17 years, n=72, 53, 51, 85 | 2 | 2 | 4 | 7

6. Secondary Outcome: Number of Participants Sustained Photophobia-free From 2-24 Hours
Description: Participants with sustained freedom from photophobia were those with an absence of photophobia (sensitivity to light) from 2 to 24 hours post-dose without the use of rescue medication.
Time Frame: 2 to 24 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 144 | 96 | 96 | 151
participants
  Total Population, n=144, 96, 96, 151 | 44 | 48 | 43 | 75
  12-14 years, n=71, 43, 46, 65 | 25 | 21 | 21 | 35
  15-17 years, n=73, 53, 50, 86 | 19 | 27 | 22 | 40

7. Secondary Outcome: Number of Participants Sustained Phonophobia-free From 2-24 Hours
Description: Participants with sustained freedom from phonophobia were those with an absence of phonophobia (sensitivity to sound) from 2 to 24 hours post-dose without the use of rescue medication.
Time Frame: 2 to 24 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 144 | 96 | 96 | 151
participants
  Total Population, n=144, 96, 96, 151 | 47 | 48 | 51 | 79
  12-14 years, n=71, 43, 46, 65 | 27 | 24 | 31 | 36
  15-17 years, n=73, 53, 50, 86 | 20 | 24 | 20 | 43

8. Secondary Outcome: Number of Participants Sustained Nausea-free From 2-24 Hours
Description: Participants with sustained freedom from nausea were those with an absence of nausea from 2 to 24 hours post-dose without the use of rescue medication.
Time Frame: 2 to 24 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 144 | 95 | 96 | 151
participants
  Total Population, n=144, 95, 96, 151 | 68 | 67 | 64 | 94
  12-14 years, n=71, 43, 46, 65 | 39 | 31 | 33 | 43
  15-17 years, n=73, 52, 50, 86 | 29 | 36 | 31 | 51

9. Secondary Outcome: Number of Participants Who Used Rescue Medication From 2 to 24 Hours Post Dose
Description: Rescue medication was defined as an additional medication taken by participants for the treatment of migraine pain or associated symptoms within 24 hours of dosing with investigational product. Permitted rescue medications included oral naproxen sodium (maximum 15 mg/kg), oral over-the-counter pain reliever, and anti-emetics. This outcome measure included only participants who rescued from 2 to 24 hours post-dose, inclusive.
Time Frame: 2 to 24 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 145 | 96 | 97 | 152
participants
  Total Population, n=145, 96, 97, 152 | 47 | 14 | 16 | 21
  12-14 years, n=71, 43, 46, 65 | 21 | 5 | 6 | 10
  15-17 years, n=74, 53, 51, 87 | 26 | 9 | 10 | 11

10. Secondary Outcome: Number of Participants Who Used Their First Dose of Rescue Medication Through the Indicated Time Points
Description: Rescue medication was defined as an additional medication taken by participants for the treatment of migraine pain or associated symptoms within 24 hours of dosing with double-blind treatment. In addition to participants who rescued from 2 to 24 hours post-dose, inclusive, this outcome measure also included nine protocol violators who rescued < 2 hours post-treatment.
Time Frame: Dosing to 24 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 145 | 96 | 96 | 152
participants
  Total Population, 1 hour, n=145, 96, 96, 152 | 2 | 0 | 0 | 2
  Total Population, 2 hours, n=145, 96, 96, 152 | 10 | 0 | 6 | 3
  Total Population, 3 hours, n=145, 96, 96, 152 | 29 | 6 | 11 | 15
  Total Population, 4 hours, n=145, 96, 96, 152 | 34 | 6 | 13 | 16
  Total Population, 8 hours, n=145, 96, 96, 152 | 45 | 9 | 15 | 20
  Total Population, 12 hours, n=145, 96, 96, 152 | 48 | 11 | 15 | 20
  Total Population, 18 hours, n=145, 96, 96, 152 | 50 | 13 | 15 | 22
  Total Population, 24 hours, n=145, 96, 96, 152 | 52 | 14 | 17 | 23
  12-14 years, 1 hour, n=71, 43, 46, 65 | 1 | 0 | 0 | 0
  12-14 years, 2 hours, n=71, 43, 46, 65 | 4 | 0 | 1 | 1
  12-14 years, 3 hours, n=71, 43, 46, 65 | 11 | 1 | 2 | 7
  12-14 years, 4 hours, n=71, 43, 46, 65 | 14 | 1 | 4 | 8
  12-14 years, 8 hours, n=71, 43, 46, 65 | 20 | 4 | 4 | 10
  12-14 years, 12 hours, n=71, 43, 46, 65 | 10 | 4 | 4 | 10
  12-14 years, 18 hours, n=71, 43, 46, 65 | 21 | 4 | 4 | 10
  12-14 years, 24 hours, n=71, 43, 46, 65 | 22 | 5 | 6 | 10
  15-17 years, 1 hour, n=74, 53, 50, 87 | 1 | 0 | 0 | 2
  15-17 years, 2 hours, n=74, 53, 50, 87 | 6 | 0 | 5 | 2
  15-17 years, 3 hours, n=74, 53, 50, 87 | 18 | 5 | 9 | 8
  15-17 years, 4 hours, n=74, 53, 50, 87 | 20 | 5 | 9 | 8
  15-17 years, 8 hours, n=74, 53, 50, 87 | 25 | 5 | 11 | 10
  15-17 years, 12 hours, n=74, 53, 50, 87 | 28 | 7 | 11 | 10
  15-17 years, 18 hours, n=74, 53, 50, 87 | 29 | 9 | 11 | 12
  15-17 years, 24 hours, n=74, 53, 50, 87 | 30 | 9 | 11 | 13

11. Secondary Outcome: Number of Participants Nausea-free at 2 Hours Post-dose
Description: The number of participants who did not have nausea at 2 hours post dose was analzyed.
Time Frame: 2 hours after single dose of double-blind treatment (Randomization through Week 13)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 144 | 95 | 96 | 151
participants
  Total Population, n=144, 95, 96, 151 | 101 | 78 | 74 | 106
  12-14 years, n=71, 43, 46, 65 | 55 | 36 | 38 | 47
  15-17 years, n=73, 52, 50, 86 | 46 | 42 | 36 | 59

12. Other Pre Specified Outcome: Mean Age of Participants at Baseline Categorized by Age Group
Description: The mean age of participants at baseline was calculated for all participants in the 12 to 14 year and 15 to 17 year age groups.
Time Frame: Baseline
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Years
Groups:
- 12 to 14 Years Age Group: Participants 12 to 14 years old treated one moderate to severe migraine attack with one tablet of double-blind treatment (placebo or one of the three sumatriptan/naproxen combination groups) within a 12-week period
- 15 to 17 Years Age Group: Participants 15 to 17 years old treated one moderate to severe migraine attack with one tablet of double-blind treatment (placebo or one of the three sumatriptan/naproxen combination groups) within a 12-week period
Arm/Group | 12 to 14 Years Age Group | 15 to 17 Years Age Group
Number analyzed (Participants) | 225 | 265
Years | 13.1 (0.79) | 16.1 (0.84)

13. Other Pre Specified Outcome: Number of Participants Randomized to Double-blind Treatment in the Indicated Age Categories at Baseline
Description: The number of participants receiving double-blind treatment were reported according to age.
Time Frame: Baseline
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg
Number analyzed (Participants) | 145 | 96 | 97 | 152
Participants
  12-14 years | 71 | 43 | 46 | 65
  15-17 years | 74 | 53 | 51 | 87

14. Other Pre Specified Outcome: Number of Female and Male Participants Categorized by Age Group
Description: The gender of participants at baseline was reported for all participants in the 12 to 14 year and 15 to 17 year age groups.
Time Frame: Baseline
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | 12 to 14 Years Age Group | 15 to 17 Years Age Group
Number analyzed (Participants) | 225 | 265
Participants
  Female | 114 | 173
  Male | 111 | 92

15. Other Pre Specified Outcome: Number of Participants of the Indicated Race Categorized by Age Group
Description: The race of participants at baseline was reported for all participants in the 12 to 14 year and 15 to 17 year age groups.
Time Frame: Baseline
Population: ITT Population
Measure: Number; unit: Participants
Arm/Group | 12 to 14 Years Age Group | 15 to 17 Years Age Group
Number analyzed (Participants) | 225 | 265
Participants
  African American/African Heritage | 31 | 32
  American Indian or Alaska Native | 1 | 0
  Asian | 2 | 2
  Native Hawaiian or other Pacific Islander | 1 | 0
  White | 181 | 216
  African American/African Heritage and White | 2 | 4
  American Indian or Alaska Native and White | 4 | 4
  Asian and Native Hawaiian/other Pacific Islander | 0 | 1
  Asian and White | 2 | 3
  Native Hawaiian/ other Pacific Islander and White | 0 | 2
  Missing | 1 | 1

16. Other Pre Specified Outcome: Mean Weight of Participants at Baseline Categorized by Age Group
Description: The mean weight of participants at baseline was calculated for all participants in the 12 to 14 year and 15 to 17 year age groups.
Time Frame: Baseline
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | 12 to 14 Years Age Group | 15 to 17 Years Age Group
Number analyzed (Participants) | 225 | 265
Kilograms (kg) | 58.7 (15.55) | 69.6 (17.78)

17. Other Pre Specified Outcome: Mean Body Mass Index of Participants at Baseline Categorized by Age Group
Description: The mean body mass index of participants at baseline was calculated for all participants in the 12 to 14 year and 15 to 17 year age groups. Body mass index is calculated as: weight (kilograms [kg]) divided by height (meters [m]^2).
Time Frame: Baseline
Population: ITT Population
Measure: Mean (Standard Deviation); unit: Kilograms per meters squared (kg/m^2)
Arm/Group | 12 to 14 Years Age Group | 15 to 17 Years Age Group
Number analyzed (Participants) | 225 | 265
Kilograms per meters squared (kg/m^2) | 22.6 (5.06) | 24.6 (5.44)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and AEs were collected from the start of investigational product (IP) in the Run-In Phase until follow-up (up through 1 week after single dose of double-blind IP for participants who took double-blind IP, up to Week 26).
Description: Treatment-emergent SAEs/AEs occurring in the Double-blind Treatment Phase are shown for Arms 1-4. Single-blind placebo-emergent SAEs/AEs occurring in the Run-In Phase are shown for Arm 5.
Groups:
- Placebo: A single matching double-blind placebo tablet taken within a 12-week period
- Single-blind Run-In Phase Placebo: One tablet of single-blind placebo taken during the Run-In Phase
Arm/Group | Placebo | Sumatriptan 10 mg/ Naproxen 60 mg | Sumatriptan 30 mg/ Naproxen 180 mg | Sumatriptan 85 mg/ Naproxen 500 mg | Single-blind Run-In Phase Placebo
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/96 | 0/97 | 0/152 | 2/683
Other Adverse Events (participants affected / at risk) | 3/145 | 0/96 | 3/97 | 4/152 | 11/683
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Sumatriptan 10 mg/ Naproxen 60 mg (N=96) | Sumatriptan 30 mg/ Naproxen 180 mg (N=97) | Sumatriptan 85 mg/ Naproxen 500 mg (N=152) | Single-blind Run-In Phase Placebo (N=683)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Sumatriptan 10 mg/ Naproxen 60 mg (N=96) | Sumatriptan 30 mg/ Naproxen 180 mg (N=97) | Sumatriptan 85 mg/ Naproxen 500 mg (N=152) | Single-blind Run-In Phase Placebo (N=683)
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 1 | 10
Hot flush (Vascular disorders) | 0 | 0 | 2 | 1 | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.